CLINICAL TRIAL: NCT05673590
Title: A Phase III, Open-label, Randomized, Controlled Clinical Study of Utidelone Versus Docetaxel in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Previously Failed Platinum-containing Chemotherapy Regimens
Brief Title: Utidelone Versus Docetaxel in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG01-2101
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-12

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Keywords: Previously Failed, Platinum-Containing Chemotherapy Regimens
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The treatment group-Utidelone monotherapy (Experimental): Drug: Utidelone Injection Dose: 40 mg/m2/d intravenously Regimen: once daily on days 1-5 in a 21-day cycle
  Interventions: Drug: Utidelone Injection
- The control group-Docetaxel monotherapy (Active Comparator): Drug: Docetaxel Injection Dose:75 mg/m2/d, administered intravenously Regimen: once on day 1 in a 21-day cycle
  Interventions: Drug: Docetaxel Injection

INTERVENTIONS:
Drug: Utidelone Injection — Pretreatment: diphenhydramine 40 mg by intramuscular injection or oral administration, and dexamethasone10 mg and cimetidine 300 mg by intravenous injection 30 minutes prior to Utidelone iv drip at the first day of each cycle. The dose of dexamethasone and diphenhydramine can be halved by the physician based on patient's condition in the following day through the fifth day in each cycle, as detailed in the protocol.
  Dexamethasone 8 mg per oral, bid, one day prior to docetaxel iv drip for 3 days.
  The treatment group will be treated with Utidelone Injection at 40 mg/m2/d intravenously once daily on days 1-5 in a 21-day cycle until disease progression or an occurrence of intolerable toxicities.
  Arms: The treatment group-Utidelone monotherapy
Drug: Docetaxel Injection — Pretreatment: Dexamethasone should be administered orally for 3 days at 16 mg per day (8 mg twice daily), starting one day before the start of Docetaxel.
  The control group will be treated with Docetaxel Injection at 75 mg/m2/d, administered intravenously once on day 1. Patients in this group will be treated in 21-day cycles until disease progression or intolerable toxicities occurs.
  Arms: The control group-Docetaxel monotherapy

SUMMARY:
The purpose of this clinical trial is to compare Utidelone with Docetaxel in patients with locally advanced or metastatic non-small cell lung cancer previously failed platinum-containing chemotherapy regimens. This phase III, open-label, randomized controlled trial aims to evaluate and compare the efficacy and safety of Utidelone and Docetaxel in the aforementioned lung cancers.

DETAILED DESCRIPTION:
In this study, 612 patients will be screened, enrolled and randomly assigned in a 1:1 ratio to either the Utidelone (40 mg/m2/d intravenously once daily on days 1-5) treatment or the docetaxel (75 mg/m2/d, intravenously once on day 1) control group, stratified by prior immunotherapy status (PD-1/PD-L1 vs. no PD-1/PD-L1). Both groups will be treated in a 21-day cycle until disease progression or an occurrence of intolerable toxicities. Tumor assessments will be performed at baseline and every 6 weeks (±7 days) after randomization and continued until disease progression as assessed by RECIST v1.1 criteria, with or without discontinuation of study treatment; the EORTC QLQ-C30 questionnaire will be used to assess patients' quality of life based on a signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the informed consent form and commit to complying with the requirements of this study.
2. Male or female, ≥ 18 years of age, ≤ 70 years of age.
3. Histologically or cytologically confirmed NSCLC, diagnosed as stage IV or stage IIIB-IIIC not amenable to radical surgery according to the IASLC (International Association for the Study of Lung Cancer) 8th edition staging system.
4. The subject has at least one evaluable lesion (measurable or non-measurable) by the RECIST 1.1.
5. The subject must have received a prior systemic chemotherapy (including neoadjuvant/adjuvant therapy) with a platinum-containing regimen, and are allowed to have ≤ 2 prior lines of chemotherapy for advanced cancer (excluding neoadjuvant/adjuvant chemotherapy).
6. Patients without driver genes can be treated with/ not be treated with PD-1/PD-L1 inhibitors previously.
7. EGFR-positive patients are required to have received at least one or more EGFR-TKI (including Erlotinib, Gefitinib, Icotinib, Afatinib, Osimertinib, or other TKI for EGFR mutations, etc.), with disease progression or intolerance during or after treatment.

   * Patients having had disease progression or intolerance to Osimertinib or other third-generation EGFR-TKI are eligible for enrollment (regardless of prior treatment with first/second-generation EGFR-TKI)
   * Patients having had disease progression or intolerance to first- or second-generation EGFR-TKI (e.g., Erlotinib, Gefitinib, Icotinib, Afatinib, etc.) without evidence of EGFR T790M mutation after this treatment are eligible for enrollment.
8. ALK fusion-positive patients who have received at least one or more ALK-TKI therapies and experienced disease progression or intolerance during or after treatment.

   -Patients having had disease progression or intolerance to the third-generation ALK-TKI Lorlatinib are eligible for enrollment (regardless of prior treatment with first- or second-generation ALK-TKI).
9. Baseline routine blood tests within 1 week prior to enrollment is normal, with CTCAE grade ≤1 (based on normal values at each site's laboratory). No rhG-CSF use and no blood transfusion/EPO etc. within 14 days prior to enrollment.

   * White blood cell count (WBC) ≥4.0 × 109/L.
   * Neutrophil count (ANC) ≥ 1.5 × 109/L.
   * platelet count (PLT) ≥ 100 × 109/L
   * Hemoglobin ≥9.0 g/dL.
10. Blood biochemistry test result is normal within 1 week prior to enrollment, with CTCAE grade ≤1 (based on normal values at each site's laboratory).

    * Total bilirubin (TBIL) ≤ 1.5× the upper limit of normal value (ULN)
    * Serum Glutamic Pyruvic Transaminase/Alanine Amino transferease (SGPT /ALT) ≤ 3× ULN (in the case of liver metastases ≤ 5 × ULN)
    * Serum Glutamic-oxaloacetic Transaminase/Aspartate Aminotransferase (SGOT /AST) ≤ 3× ULN (in the case of liver metastases ≤ 5 × ULN)
    * Creatinine clearance (Ccr) ≥60 ml/min.
11. ECOG performance status 0-1.
12. Fertile males and females of childbearing potential must agree to use effective contraception during the study and within 90 days after the last dose. The blood or urine pregnancy test for female patients of childbearing age prior to enrollment must be negative.
13. Patients with a life expectancy of more than 3 months.

Exclusion Criteria:

1. Patients who had other malignancies within the past 5 years, excluding cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid cancer.
2. Patients who have received antitumor therapy, including chemotherapy, radiotherapy, biologic therapy, targeted therapy, immunotherapy, or antitumor herbal therapy, within 4 weeks or 5 half-lives (≥ 2 weeks), whichever is shorter, prior to the first dose of the study drug.
3. Patients who have had surgery of their major organs (excluding puncture biopsy) or had major injuries within 4 weeks prior to the first dose of study drug, or require elective surgery during the study.
4. Patients with symptomatic peripheral neuropathy with CTCAE 5.0 grade ≥2
5. Patients with known allergic reactions to any ingredient of the study drug.
6. Patients who have previously been treated with docetaxel.
7. Patients who are pregnant (positive result from the pregnancy test) or lactating.
8. Patients whose prior adverse reactions to anti-tumor therapy have not recovered to CTCAE 5.0 grade ≤1 (except for toxicity such as alopecia which poses no safety risk in the judgment of the investigator).
9. Patients with symptomatic CNS metastases or meningeal metastases, or uncontrollable metastases, i.e., metastatic lesion progression confirmed by examination within 2 months after radiotherapy or other localized treatment, or those who are unsuitable for enrollment in the judgment of the investigator.
10. Patients with uncontrollable bone metastases, i.e., patients who have had fracture or have the risk of fracture in recent days, patients who need surgery or localized radiotherapy in recent days, and patients under critical conditions in the judgment of the investigator.
11. Patients with uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently)
12. Patients with an active infection that currently requires systemic anti-infective therapy
13. Patients having a history of immunodeficiency, including a positive HIV antibody test.
14. Patients with active hepatitis B/C infection; patients with known active infection of syphilis.
15. Patients with history of severe cardiovascular disease, including but not limited to:

    * Serious cardiac rhythm or conduction abnormalities such as ventricular arrhythmias requiring clinical intervention, second- to third- degree atrioventricular block; mean QTcF >470ms from 3 12-lead ECGs at rest.
    * Patients who had acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular events at Class 3 or higher within 6 months prior to the first dose.
    * Patients with clinically uncontrollable hypertension.
    * Patients with other high-risk cardiac conditions in the judgment of the investigator.
16. Patients with uncontrolled diabetes mellitus.
17. Patients with mental disorders or poor compliance.
18. Patients who concurrently participate in another clinical trial or use another investigational treatment.
19. Subjects who, in the opinion of the investigator, have a history of other serious systemic diseases, or other reasons that make participation in this trial inadvisable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 36 months
  Comparing the OS of Utidelone and Docetaxel for locally advanced or metastatic non-small cell lung cancer patients who previously failed Platinum-containing chemotherapy regimens

SECONDARY OUTCOMES:
Progression Free Survival | 36 months
  Imaging-provable disease progression
Objective Response Rate | 36 months
  The number of patients with an observed best efficacy rating of CR or PR as a percentage of the total number of evaluable patients according to RECIST 1.1.
Clinical Benefit Rate | 36 months
  The number of patients with best efficacy ratings of CR, PR and SD as a percentage of the total number of evaluable patients according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China